CLINICAL TRIAL: NCT01032187
Title: Efficacy and Safety of Amphotericin B Deoxycholate Compared to Meglumine Antimoniate for Treatment of Visceral Leishmaniasis in Brazilian Children
Brief Title: Amphotericin B to Treat Visceral Leishmaniasis in Brazilian Children
Acronym: LVTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Gustavo Adolfo Sierra Romero, Associate Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVTO-I
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; Amphotericin B deoxycholate; Meglumine antimoniate; Children; Brazil
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Meglumine Antimoniate; amphotericin B, deoxycholate drug combination; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meglumine antimoniate (Active Comparator): 20mg/kg/day IV for 20 days
  Interventions: Drug: Meglumine antimoniate
- Anfo B (Experimental): Amphotericin B-deoxycholate, 1mg/kg/day IV for 14 days
  Interventions: Drug: Amphotericin B-deoxycholate

INTERVENTIONS:
Drug: Meglumine antimoniate — 20mg/kg/day IV for 20 days
  Other Names: Glucantime
  Arms: Meglumine antimoniate
Drug: Amphotericin B-deoxycholate — Amphotericin B-deoxycholate 1 mg/kg/day IV for 14 days
  Other Names: Fungizone
  Arms: Anfo B

SUMMARY:
The purpose of this study is to determine if amphotericin B is effective against visceral leishmaniasis in Brazilian children. Amphotericin B will be compared to meglumine antimoniate which is the current approved drug used for this disease in Brazil.

DETAILED DESCRIPTION:
Despite their high toxicity, antimonials and amphotericin B deoxycholate are commonly used for treating visceral leishmaniasis (VL). Few studies showing conflictive data about their efficacy and adverse events in pediatric population are available. This study aimed to evaluate efficacy and safety of amphotericin B deoxycholate vs. that of N-methylglucamine antimoniate in treating pediatric VL in Brazil. This was a randomized, open-label, 2-arm and controlled pilot clinical trial. Treatment naïve children and adolescents with VL without signs of severe illness were treated with N-methylglucamine antimoniate or amphotericin B deoxycholate. All patients were diagnosed with positive direct examination and/or positive PCR for Leishmania spp. performed in bone marrow samples. The primary efficacy end-point was VL cure determined after 180 days of completion of treatment. The analysis was performed using intention-to-treat (ITT) and per protocol (PP) analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of visceral leishmaniasis: fever plus hepatomegaly or splenomegaly
* Diagnosis of visceral leishmaniasis confirmed through parasite visualization in bone marrow smears or positive serology (indirect immunofluorescent antibody test or rK39 rapid test)or positive kDNA PCR test

Exclusion Criteria:

* Any of the following laboratory findings

  * Total serum bilirubin higher than 2,5 mg/dL
  * Serum SGOT higher than 5 times the upper normal level
  * Serum SGPT higher than 5 times the upper normal level
  * Prothrombin time concentration lower than 70%
  * Abnormal serum creatinine
* Any of the following signs or symptoms

  * Generalized edema
  * Severe malnutrition
  * Systemic inflammatory response syndrome
* Any of the following conditions

  * HIV infection/disease
  * Diabetes
  * Corticoid or immunosuppressive drugs use
  * Symptomatic heart diseases
  * Chronic hepatic or renal diseases
  * Lupus erythematosus

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cure rate | 3 months

SECONDARY OUTCOMES:
Improvement rate | 30 days
Adverse events rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Myrlena RM Borges, MsC, Principal Investigator — Federal University of Tocantins; Gustavo AS Romero, PhD, Study Chair — University of Brasilia
Locations (2):
- Brazil (2):
  - Hospital de Doenças Tropicais, Araguaína, Tocantins
  - Hospital Dona Regina, Palmas, Tocantins

REFERENCES:
- [Result] Borges MM, Pranchevicius MC, Noronha EF, Romero GA, Carranza-Tamayo CO. Efficacy and safety of amphotericin B deoxycholate versus N-methylglucamine antimoniate in pediatric visceral leishmaniasis: an open-label, randomized, and controlled pilot trial in Brazil. Rev Soc Bras Med Trop. 2017 Jan-Feb;50(1):67-74. doi: 10.1590/0037-8682-0455-2016. PMID 28327804